CLINICAL TRIAL: NCT03532399
Title: Pharmacokinetics of Bivalirudin for Pediatric Anticoagulation
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Katherine Zaleski, Instructor in Anaesthesia, Boston Children's Hospital
Other Study IDs: IRB-P00027930
Record Dates: First submitted 2018-04-17; First posted 2018-05-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Drug Effect
Keywords: Bivalirudin
MeSH Terms: interventions — bivalirudin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Pediatric Cardiac Catheterization
  Interventions: Drug: Bivalirudin
- Pediatric Cardiac Surgery
  Interventions: Drug: Bivalirudin
- Pediatric Extracorporeal Life Support (ECLS)
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Bivalirudin — CPB: Per hospital protocol, bivalirudin 1 mg/kg IV will be administered to the patient 10 minutes prior to the start of CPB along with an infusion of bivalirudin at 2.5 mg/kg/hr. Additional bolus doses of 0.5 to 1 mg/kg will be administered for ACTs less than the specified target (either 2 times baseline ACT or > 400 seconds per the discretion of the patient's providers). 50mg of bivalirudin will be administered to the bypass circuit.
  Cardiac Catheterization: Bivalirudin will be administered to the patient as 0.75mg/kg IV bolus followed by a 1.75mg/kg/hr infusion for the length of the procedure. Changes in infusion rate or bolus dosing during the procedure and post-procedure will be at the discretion of the patient's care providers.
  ECMO/VAD: Dosing will be informed by the hospital's formulary recommendations(http://online.lexi.com/lco/action/doc/retrieve/docid/chibos_f/6317841), but will ultimately be determined by patient's primary provider.

SUMMARY:
This study will measure plasma concentrations of bivalirudin in pediatric patients undergoing cardiac catheterization, cardiac surgical procedures utilizing cardiopulmonary bypass (CPB), or extracorporeal support with ECMO, ventricular support devices (VAD) or lung-assist devices (LAD). The aim is to understand the pharmacokinetics of bivalirudin in these settings.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patient (age less than 18 years)
* weight > 3kg
* scheduled to undergo 1) cardiac catheterization, 2)cardiac surgical procedure utilizing CPB, and/or 3) the institution of extracorporeal support
* must already require the administration of bivalirudin as part of their treatment plan

Exclusion Criteria:

* Age equal to or greater than 18 years,
* weight less than 3kg
* end-stage renal failure requiring renal replacement therapy.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric (age less than 18 years and more than 3kg) patients who present to Boston Children's Hospital (BCH) for cardiac catheterization, a cardiac surgical procedure utilizing CPB, or the institution of extracorporeal support and who require the administration of bivalirudin as part of their treatment plan will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Plasma Bivalirudin Concentration | Throughout the duration of treatment with bivalirudin and for one hour after the infusion is stopped. To be specific: 1. In CPB and cath lab cases arm: average 6 hours. 2. In ECLS arm: average 10 days.
  The primary end-point will be the plasma bivalirudin concentration (nanogram/mL) measured at multiple set time-points throughout the administration of bivalirudin in order to delineate the pharmacokinetic profile in the pediatric population.

SECONDARY OUTCOMES:
thrombotic complications | Data will be assessed continuously in the procedural groups throughout the duration of the infusion and then continued weekly throughout the length of the hospital stay up to one year from enrollment.
  arterial, venous, and/or CPB/ECMO/VAD thrombosis; embolic stroke
bleeding in excess of expectations for a given procedure or ECLS modality | Data will be assessed continuously in the procedural groups throughout the duration of the infusion and then continued weekly throughout the length of the hospital stay up to one year from enrollment.
mortality | Data will be assessed continuously in the procedural groups throughout the duration of the infusion and then continued weekly throughout the length of the hospital stay or until death up to one year from enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No